CLINICAL TRIAL: NCT01785563
Title: Nasal Noninvasive NAVA Provides Ventilation in the Very Low Birth Weight Infant
Brief Title: Nasal Noninvasive NAVA in the Very Low Birth Weight Infant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarah T Colaizy (Other)
Responsible Party: Sponsor-Investigator, Tarah T Colaizy, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201208771
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Results first posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Inadequate; Pulmonary Ventilation, Newborn; Infant, Very Low Birth Weight
Keywords: NAVA; NIV-NAVA; VLBW; electrical activity of the diaphragm; neural trigger, mechanical ventilation; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Nasal NIV-NAVA (Experimental): Infants will be transitioned from their current mode of ventilation to nasal NIV-NAVA. If patients are currently on nasal NIV-NAVA an increase in the NAVA level will be utilized for the intervention.
  Interventions: Device: Nasal NIV-NAVA

INTERVENTIONS:
Device: Nasal NIV-NAVA — Infants will be placed on nasal NIV-NAVA. Patients initial NAVA level will be set to generate a peak inspiratory pressure that is 8 cm of water greater than their current peak end expiratory pressure. If the infants are on nasal NIV-NAVA at the time of study entry their NAVA level will be increased by 50% rounded up to the nearest 0.1 cm of water per microvolt.
  Other Names: noninvasive; neurally adjusted ventilatory assist; nasal pharyngeal

SUMMARY:
The purpose of this study is to determine if a new type of mechanical ventilation, or breathing machine (called neurally adjusted ventilatory assist or NAVA), will provide additional support to infants who were born prematurely. Investigators are looking to determine if in two hours infants who weighed less than 1500 grams or 3 pounds 5 ounces, will demonstrate a decrease in the amount of carbon dioxide (the gas that humans exhale) dissolved in their blood as compared to prior to starting the study. This will be accomplished by enrolling infants who are stable on their current type of mechanical breathing that provides a constant air flow into the infant. This type of mechanical support helps keep the lungs inflated but does not help remove carbon dioxide. This study will change the type of mechanical support to a type of support called neurally adjusted ventilatory assist or NAVA. This type of mechanical support detects when the infant is breathing in by having electrical sensors on a feeding tube that is placed into the stomach through the nose or mouth. These electrical sensors detect when the diaphragm or the muscle that helps humans breath is trying to take a breath in. When the NAVA ventilator senses the attempt to breath, it provides additional air flow to make the effort of breathing easier. The ventilator will be attached to a tube or cannula that is placed into the infant's nose. After two hours of being on the NAVA ventilator a repeat measure of carbon dioxide in the blood will be performed by taking a small amount of blood from the infant's heel.

DETAILED DESCRIPTION:
Baseline Data Collection:

Demographic data: Patient gestational age at delivery, maternal betamethasone therapy, APGAR scores, admission weight, receipt of surfactant administered, age at extubation, time since extubation, current post menstrual age, and current weight.

Baseline vitals and ventilation mode: Heart rate, blood pressure, FiO2 (fraction of inspired oxygen), oxygen saturations, transcutaneous partial pressure of carbon dioxide (TCO2) and current mode of ventilation will be recorded four times in a one minute period and the values average to minimize normal variation. Intervention time will be manipulated to begin no later than one hour after the previous feeding, as to minimize interruption of feedings to no greater than 30 minutes.

Safety Safety: TCO2 monitor will be attached to the infant and the device will be calibrated according to protocol (reference TCO2 monitor manual). Carbon dioxide diffusion through the skin will be monitored continuously during the intervention (Bromley 08) to avoid periods of hypo or hypercarbia.

Edi (electrical activity of the diaphragm) Catheter placement: Edi catheter size will be selected according to infant's weight and length. It will be inserted according to manufacturer's guidelines and adjustments will be made to optimize positioning (reference NAVA manual).

NAVA settings:

Infants will be maintained on previous level of PEEP (positive end expiratory pressure) or calculated PEEP, rounding up to whole numbers. Initial NAVA level will be determined by starting with an initial NAVA level of 0.5 microvolts/cm of H20. The NAVA level will then be adjusted either by increasing or decreasing to generate a PIP that is a minimum of 8 cm of H2O greater than the current PEEP. Apnea alarm will be set at 5 seconds, which will initiate the NAVA back up setting if no electrical activity is detected by the Edi catheter. Back up NAVA settings will be set with a PIP of 12 cm of H20 greater than current PEEP, respiratory rate of 60 breaths per minute (RR) and inspiratory time of 0.5 seconds. Fraction of inspired oxygen (FiO2) will be adjusted to keep infant's oxygen saturations within previously established clinical parameters.

Study Intervention Procedure and Data Collection:

At initiation of intervention, and at time 30, 60, 90, and 120 minutes, heart rate (HR), respiratory rate (RR), tidal volume (TV), minute ventilation, FiO2, oxygen saturations, peak Edi and PIP will be recorded four times in a one minute period and the values average to minimize normal variation. Current NAVA settings, TCO2, and blood pressure (BP) will also be recorded. At 60 minutes of intervention if the TCO2 level has not decreased by 5 torr from baseline or has risen, the current NAVA level will be increased by 50%. At 90 minutes if the TCO2 level has not decreased by 5 torr from baseline or has risen; the NAVA level will be increased by 50% from the current level. At the completion of the study (120 minutes or pCO2 outside of established limits) the HR, RR, BP, TV, minute ventilation, FiO2, oxygen saturations, peak Edi and PIP will be recorded four times in a one minute period and the values average to minimize normal variation. A capillary blood gas will be obtained according to standard unit protocol with a warmed heel.

ELIGIBILITY:
Inclusion Criteria:

* birth weight less than 1,500 grams
* Clinical history of respiratory distress syndrome treated with surfactant
* Chronological age greater than or equal to seven days
* 48 hours post-extubation or greater
* Medically stable per primary medical team
* Receiving ventilatory support on one of the following systems via nasal pharyngeal tube or nasal prongs:continuous positive airway pressure (CPAP), intermittent mechanical ventilation (IMV), or neutrally adjusted ventilatory assistance (NAVA)
* Receiving ventilatory support via high flow nasal cannula if the flow is large enough to provide a positive end expiratory pressure (PEEP) of 6 as defined by PEEP of 6 = 0.68 * weight (kg) + 0.92
* Capillary blood gas via heel stick within 24 hours that demonstrates a pH of less than or equal to 7.35 and/or a partial pressure of carbon dioxide (pCO2) greater than or equal to 45 mmHg

Exclusion criteria:

* Severe congenital abnormalities
* Grade III or IV interventricular hemorrhage.

Ages: 7 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarah T Colaizy, M.D., MPH, Principal Investigator — University of Iowa; Gary J Kummet, M.D., Study Director — University of Iowa; Jonathan C Klein, M.D., Study Director — University of Iowa
Locations (2):
- United States (2):
  - Children's Hospital of Iowa NICU, Iowa City, Iowa
  - University of Iowa, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breatnach C, Conlon NP, Stack M, Healy M, O'Hare BP. A prospective crossover comparison of neurally adjusted ventilatory assist and pressure-support ventilation in a pediatric and neonatal intensive care unit population. Pediatr Crit Care Med. 2010 Jan;11(1):7-11. doi: 10.1097/PCC.0b013e3181b0630f. PMID 19593246
- [Background] de la Oliva P, Schuffelmann C, Gomez-Zamora A, Villar J, Kacmarek RM. Asynchrony, neural drive, ventilatory variability and COMFORT: NAVA versus pressure support in pediatric patients. A non-randomized cross-over trial. Intensive Care Med. 2012 May;38(5):838-46. doi: 10.1007/s00134-012-2535-y. Epub 2012 Apr 6. PMID 22481227
- [Background] Clement KC, Thurman TL, Holt SJ, Heulitt MJ. Neurally triggered breaths reduce trigger delay and improve ventilator response times in ventilated infants with bronchiolitis. Intensive Care Med. 2011 Nov;37(11):1826-32. doi: 10.1007/s00134-011-2352-8. Epub 2011 Sep 23. PMID 21946913
- [Background] Alander M, Peltoniemi O, Pokka T, Kontiokari T. Comparison of pressure-, flow-, and NAVA-triggering in pediatric and neonatal ventilatory care. Pediatr Pulmonol. 2012 Jan;47(1):76-83. doi: 10.1002/ppul.21519. Epub 2011 Aug 9. PMID 21830318
- [Background] Bordessoule A, Emeriaud G, Morneau S, Jouvet P, Beck J. Neurally adjusted ventilatory assist improves patient-ventilator interaction in infants as compared with conventional ventilation. Pediatr Res. 2012 Aug;72(2):194-202. doi: 10.1038/pr.2012.64. PMID 22580718
- [Background] Bengtsson JA, Edberg KE. Neurally adjusted ventilatory assist in children: an observational study. Pediatr Crit Care Med. 2010 Mar;11(2):253-7. doi: 10.1097/PCC.0b013e3181b0655e. PMID 19593241
- [Background] Lee J, Kim HS, Sohn JA, Lee JA, Choi CW, Kim EK, Kim BI, Choi JH. Randomized crossover study of neurally adjusted ventilatory assist in preterm infants. J Pediatr. 2012 Nov;161(5):808-13. doi: 10.1016/j.jpeds.2012.04.040. Epub 2012 Jun 1. PMID 22658785
- [Background] Keszler M. State of the art in conventional mechanical ventilation. J Perinatol. 2009 Apr;29(4):262-75. doi: 10.1038/jp.2009.11. Epub 2009 Feb 26. PMID 19242486
- [Background] Stein H, Howard D. Neurally adjusted ventilatory assist in neonates weighing <1500 grams: a retrospective analysis. J Pediatr. 2012 May;160(5):786-9.e1. doi: 10.1016/j.jpeds.2011.10.014. Epub 2011 Dec 3. PMID 22137670
- [Background] Stein H, Firestone K, Rimensberger PC. Synchronized mechanical ventilation using electrical activity of the diaphragm in neonates. Clin Perinatol. 2012 Sep;39(3):525-42. doi: 10.1016/j.clp.2012.06.004. PMID 22954267
- [Background] Beck J, Reilly M, Grasselli G, Mirabella L, Slutsky AS, Dunn MS, Sinderby C. Patient-ventilator interaction during neurally adjusted ventilatory assist in low birth weight infants. Pediatr Res. 2009 Jun;65(6):663-8. doi: 10.1203/PDR.0b013e31819e72ab. PMID 19218884
- [Background] Beck J, Brander L, Slutsky AS, Reilly MC, Dunn MS, Sinderby C. Non-invasive neurally adjusted ventilatory assist in rabbits with acute lung injury. Intensive Care Med. 2008 Feb;34(2):316-23. doi: 10.1007/s00134-007-0882-x. Epub 2007 Oct 25. PMID 17960364
- [Background] Bertrand PM, Futier E, Coisel Y, Matecki S, Jaber S, Constantin JM. Neurally adjusted ventilatory assist vs pressure support ventilation for noninvasive ventilation during acute respiratory failure: a crossover physiologic study. Chest. 2013 Jan;143(1):30-36. doi: 10.1378/chest.12-0424. PMID 22661448
- [Background] Cammarota G, Olivieri C, Costa R, Vaschetto R, Colombo D, Turucz E, Longhini F, Della Corte F, Conti G, Navalesi P. Noninvasive ventilation through a helmet in postextubation hypoxemic patients: physiologic comparison between neurally adjusted ventilatory assist and pressure support ventilation. Intensive Care Med. 2011 Dec;37(12):1943-50. doi: 10.1007/s00134-011-2382-2. Epub 2011 Oct 18. PMID 22005826
- [Background] Piquilloud L, Tassaux D, Bialais E, Lambermont B, Sottiaux T, Roeseler J, Laterre PF, Jolliet P, Revelly JP. Neurally adjusted ventilatory assist (NAVA) improves patient-ventilator interaction during non-invasive ventilation delivered by face mask. Intensive Care Med. 2012 Oct;38(10):1624-31. doi: 10.1007/s00134-012-2626-9. Epub 2012 Aug 3. PMID 22885649
- [Background] Schmidt M, Dres M, Raux M, Deslandes-Boutmy E, Kindler F, Mayaux J, Similowski T, Demoule A. Neurally adjusted ventilatory assist improves patient-ventilator interaction during postextubation prophylactic noninvasive ventilation. Crit Care Med. 2012 Jun;40(6):1738-44. doi: 10.1097/CCM.0b013e3182451f77. PMID 22610179

RESULTS

PARTICIPANT FLOW:
Groups:
- Nasal Non-Invasive NAVA Group: Infants < 1500g birthweight, who were intubated and received surfactant at birth, at least 7 days old, and at least 48 hours after endotracheal extubation. Infants must be receiving respiratory support at study entry, including CPAP or non-invasive mechanical ventilation.
Period: Overall Study
Arm/Group | Nasal Non-Invasive NAVA Group
Started | 40
Completed | 27
Not Completed | 13
Not completed — Physician Decision | 10
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nasal Non-Invasive NAVA Group
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 47 (29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 19
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27
screening capillary blood gas pH [Mean (Full Range); unit: ph units] | 7.38 [7.3 to 7.48]

OUTCOME MEASURES:

1. Primary Outcome: Change in Partial Pressure of Carbon Dioxide on Capillary Blood Gas
Description: difference between pCO2 (mm Hg) on capillary blood gas obtained within 6 hours of study and immediately after 2 hour study period
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nasal Non-Invasive NAVA Group
Number analyzed (Participants) | 27
mm Hg | 0.019 (0.037)

2. Secondary Outcome: Change in Fraction of Inspired Oxygen
Description: difference between fiO2 at start of study and that at the last measurement timepoint at 120 minutes
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: percentage of oxygen in inspired gas
Arm/Group | Nasal Non-Invasive NAVA Group
Number analyzed (Participants) | 27
percentage of oxygen in inspired gas | -0.012 (0.0463)

ADVERSE EVENTS:
Time Frame: Each subject was monitored for adverse events potentially attributable to the study intervention from the time of enrollment and completion of the study until their discharge from the hospital, which varied from 3 weeks to 3 months.
Arm/Group | Nasal Non-Invasive NAVA Group
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT01785563/Prot_SAP_000.pdf